CLINICAL TRIAL: NCT00244712
Title: A 96-Week, Phase IV, Randomized, Double-Blind, Multicenter Study of the Safety and Efficacy of EPZICOM Versus TRUVADA Administered in Combination With KALETRA in Antiretroviral-Naive HIV-1 Infected Subjects
Brief Title: Abacavir/Lamivudine Versus Emtricitabine/Tenofovir Both In Combination With Lopinavir/Ritonavir For The Treatment Of HIV
Acronym: HEAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPZ104057; EPZ104057
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Results first posted 2009-09-15 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-06

CONDITIONS: HIV Infection
Keywords: HEAT; Antiretroviral-naive; HIV; EPZICOM; TRUVADA; KALETRA; once-daily
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; abacavir, lamivudine drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- ABC/3TC (Experimental): The intervention is a regimen containing abacavir/lamivudine + tenofovir/emtricitabine placebo +lopinavir/ritonavir.
  Interventions: Drug: abacavir/lamivudine
- TDF/FTC (Active Comparator): The intervention is a regimen containing tenofovir/emtricitabine + abacavir/lamivudine placebo + lopinavir/ritonavir.
  Interventions: Drug: emtricitabine/tenofovir

INTERVENTIONS:
Drug: emtricitabine/tenofovir — The intervention is an active comparator regimen containing tenofovir/emtricitabine + abacavir/lamivudine placebo + lopinavir/ritonavir.
  Arms: TDF/FTC
Drug: abacavir/lamivudine — The experimental intervention is a regimen containing abacavir/lamivudine + tenofovir/emtricitabine placebo + lopinavir/ritonavir.
  Arms: ABC/3TC

SUMMARY:
This study was designed to test the safety and effectiveness of EPZICOM(abacavir/lamivudine) and TRUVADA (emtricitabine/tenofovir) for the treatment of HIV infection when both are used in combination with KALETRA (lopinavir/ritonavir) over 96 weeks

ELIGIBILITY:
Inclusion criteria:

* Males as females at least 18 years old. (A female is eligible to enter and participate in this study if she is of: non child-bearing potential, child bearing potential with a negative pregnancy test and agrees to approved contraception methods, or agreement for complete abstinence.)
* Subject is antiretroviral-naïve (defined as having ≤14 days of prior therapy with any NRTI and no prior therapy with either a PI or NNRTI).
* Subject has plasma HIV-1 RNA ≥ 1,000 copies/mL at screening.
* Subject is willing and able to understand and provide written informed consent prior to participation in this study.

Exclusion criteria:

* Subject has an active or acute CDC Clinical Category C event (exclusive of cutaneous Kaposi's sarcoma) at screening. Treatment for the acute event must have been completed at least 30 days prior to screening.
* Subject is enrolled in one or more investigational drug protocols, which may impact HIV-1 RNA suppression.
* Subject is, in the opinion of the investigator, unable to complete the 96-week dosing period and protocol evaluations and assessments.
* Subject is either pregnant or breastfeeding.
* Subject has an ongoing clinically relevant pancreatitis or clinically relevant hepatitis at screening.
* Subject suffers from a serious medical condition, such as cirrhosis, diabetes, congestive heart failure, cardiomyopathy or other cardiac dysfunction, which in the opinion of the investigator would compromise the safety of the subject.
* Subject has a pre-existing mental, physical, or substance abuse disorder which, in the opinion of the investigator, may interfere with the subject's ability to comply with the dosing schedule and protocol evaluations and assessments.
* Subject has a history of inflammatory bowel disease or malignancy, intestinal ischemia, malabsorption, or other gastrointestinal dysfunction which may interfere with drug absorption or render the subject unable to take oral medication.
* Subject has any acute laboratory abnormality at screening, which, in the opinion of the investigator, precludes the subject's participation in the study of an investigational compound. Any grade 4 laboratory abnormality will exclude a subject from study participation.
* Subject has estimated creatinine clearance <50 mL/min via Cockroft-Gault method.
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >5 times the upper limit of normal (ULN).
* Subject has required treatment with radiation therapy or cytotoxic chemotherapeutic agents within 28 days prior to screening, or has an anticipated need for these agents within the study period.
* Subject requires treatment with immunomodulating agents (such as systemic corticosteroids, interleukins, vaccines, or interferons) within 28 days prior to Screen, or subject has received an HIV-1 immunotherapeutic vaccine within 90 days prior to Screen. Asthmatic subjects using inhaled corticosteroids are eligible for enrollment.
* Subject requires treatment with foscarnet, hydroxyurea or other agents with documented activity against HIV-1 in vitro within 28 days of study administration.
* Subjects who require treatment with the prohibited medications within 28 days of commencement of investigational product, or an anticipated need during the study.
* Subject has a history of allergy to any of the study drugs or any excipients therein

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 688 (Actual)
Dates: Start 2005-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (57):
- United States (55):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Garden Grove, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Glastonbury, Connecticut
  - GSK Investigational Site, Norwalk, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Key West, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Port Saint Lucie, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Maywood, Illinois
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Hillsborough, New Jersey
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Somers Point, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, West Reading, Pennsylvania
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Harlingen, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Longview, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Annandale, Virginia
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Hampton, Virginia
  - GSK Investigational Site, Lynchburg, Virginia
  - GSK Investigational Site, Milwaukee, Wisconsin
- Puerto Rico (2):
  - GSK Investigational Site, Ponce
  - GSK Investigational Site, San Juan

REFERENCES:
- [Derived] Smith KY, Patel P, Fine D, Bellos N, Sloan L, Lackey P, Kumar PN, Sutherland-Phillips DH, Vavro C, Yau L, Wannamaker P, Shaefer MS; HEAT Study Team. Randomized, double-blind, placebo-matched, multicenter trial of abacavir/lamivudine or tenofovir/emtricitabine with lopinavir/ritonavir for initial HIV treatment. AIDS. 2009 Jul 31;23(12):1547-56. doi: 10.1097/QAD.0b013e32832cbcc2. PMID 19542866

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 76 study sites in the US and 2 study sites in Puerto Rico between 26 July 2005 and 16 June 2006.
Pre-assignment Details: After screening, participants who had never received treatment for HIV-1 infection and had a viral load greater than or equal to 1,000 copies per milliliter of blood and any amount of CD4+ T-cells were equally randomized to 1 of 2 treatment groups.
Groups:
- Abacavir/Lamivudine (ABC/3TC) + Lopinavir/Ritonavir (LPV/RTV): 1 tablet (600mg/300mg) ABC/3TC + 800mg/200mg LPV/RTV combination therapy once daily
- Tenofovir/Emtricitabine (TDF/FTC) + LPV/RTV: 1 tablet (300mg/200mg) TDF/FTC + 800mg/200mg LPV/RTV combination therapy once daily
Period: Overall Study
Arm/Group | Abacavir/Lamivudine (ABC/3TC) + Lopinavir/Ritonavir (LPV/RTV) | Tenofovir/Emtricitabine (TDF/FTC) + LPV/RTV
Started | 343 | 345
Completed | 234 | 221
Not Completed | 109 | 124
Not completed — Adverse Event | 20 | 21
Not completed — Protocol-Defined Virologic Failure | 8 | 6
Not completed — Lack of Compliance | 10 | 11
Not completed — Lost to Follow-up | 45 | 52
Not completed — Withdrawal by Subject | 13 | 23
Not completed — Protocol Violation, disease progression | 13 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abacavir/Lamivudine (ABC/3TC) + Lopinavir/Ritonavir (LPV/RTV) | Tenofovir/Emtricitabine (TDF/FTC) + LPV/RTV | Total
Number analyzed (Participants) | 343 | 345 | 688
Age Continuous [Mean (Standard Deviation); unit: years] | 38.0 (9.80) | 38.7 (9.55) | 38.3 (9.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 69 | 125
  Male | 287 | 276 | 563
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 122 | 124 | 246
  American Indian or Alaskan Native | 0 | 1 | 1
  Asian | 6 | 9 | 15
  White | 177 | 174 | 351
  Mixed Race | 2 | 1 | 3
  Unspecified | 36 | 36 | 72
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 73 | 62 | 135
  Not Hispanic or Latino | 270 | 282 | 552
  Missing Information | 0 | 1 | 1
Baseline CD4+ Cell Count Level [Number; unit: participants]
  <50 cells per cmm | 61 | 70 | 131
  50 - <200 cells per cmm | 99 | 110 | 209
  >= 200 cells per cmm | 183 | 165 | 348
Baseline HIV-1 RNA Level [Number; unit: participants]
  <100,000 copies/mL | 188 | 205 | 393
  100,000 - <250,000 copies/mL | 68 | 75 | 143
  250,000 - <500,000 copies/mL | 37 | 33 | 70
  >=500,000 copies/mL | 50 | 32 | 82
Centers for Disease Control (CDC) Classification [Number; unit: participants] — HIV, Human Immunodeficiency Virus; AIDS, Acquired Immunodeficiency Syndrome
  participants
    A: Asymptomatic HIV infection | 229 | 240 | 469
    B: Symptomatic HIV infection | 59 | 48 | 107
    C: AIDS | 55 | 57 | 112
Hepatitis B Infection [Number; unit: participants]
  Reactive | 19 | 9 | 28
  Non-Reactive | 324 | 334 | 658
  Missing | 0 | 2 | 2
Hepatitis C Infection [Number; unit: participants]
  Reactive | 27 | 24 | 51
  Non-Reactive | 316 | 319 | 635
  Missing | 0 | 2 | 2
Baseline CD4+ Cell Count [Median (Full Range); unit: cells per cmm] | 214 [19 to 962] | 193 [19 to 953] | 202 [19 to 962]
Baseline HIV-1 RNA [Median (Full Range); unit: log10 copies/mL] — HIV-1 RNA, Human Immunodeficiency Virus type 1 Ribonucleic acid
  log10 copies/mL | 4.903 [2.658 to 6.994] | 4.844 [1.690 to 6.565] | 4.876 [1.690 to 6.994]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies/mL at Week 48 by Missing=Failure (M=F), Switched Included Analysis.
Description: A blood sample was drawn to determine the amount of HIV-1 RNA virus in copies/mL at Week 48. The percentage of participants with HIV-1 RNA <50 copies/mL were tabulated by treatment arm with stratification by baseline HIV-1 RNA (<100,000 copies/mL and >=100,000 copies/mL).
Time Frame: Week 48
Population: The Intent-To-Treat-Exposed (ITT-E) population which included all randomized participants that had received at least one dose of study medication. In the missing=failure, switched included analysis, participants who had switched their randomized treatment for other treatment were considered as failures, i.e., HIV-1 RNA >=50 copies/mL.
Measure: Number; unit: percentage of participants
Arm/Group | Abacavir/Lamivudine (ABC/3TC) + Lopinavir/Ritonavir (LPV/RTV) | Tenofovir/Emtricitabine (TDF/FTC) + LPV/RTV
Number analyzed (Participants) | 343 | 345
percentage of participants | 67.5 | 67.2
Statistical Analysis 1: Comparison: Abacavir/Lamivudine (ABC/3TC) + Lopinavir/Ritonavir (LPV/RTV) vs Tenofovir/Emtricitabine (TDF/FTC) + LPV/RTV; Test type: Non-Inferiority or Equivalence — Non-inferiority of the ABC/3TC to the TDF/FTC would be declared if the lower limit of the 2-sided 95% confidence interval on the difference in the percentage of participants with HIV-1 RNA <50 copies/mL at Week 48 [ABC/3TC minus TDF/FTC] was -12% or greater; p = 0.913, Cochran-Mantel-Haenszel; difference in response percentage = 0.39, 95% CI [-6.63 to 7.40] — Difference in response percentage = percentage in Arm 1 minus percentage in Arm 2

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies/mL at Week 48
Description: A blood sample was drawn to determine the amount of HIV-1 RNA virus in copies/mL at Week 48. The percentage of participants with HIV-1 RNA <50 copies/mL at Week 48 were tabulated by treatment arm with stratification by baseline HIV-1 RNA levels (<100,000 copies/mL and >=100,000 copies/mL).
Time Frame: Week 48
Population: The Intent-To-Treat-Exposed (ITT-E) population which included all patients that had received at least one dose of study medication. The secondary analysis methods were time to loss of virologic response (TLOVR), Observed (Obs), and missing/discontinuation=failure (M/D=F) analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Abacavir/Lamivudine (ABC/3TC) + Lopinavir/Ritonavir (LPV/RTV) | Tenofovir/Emtricitabine (TDF/FTC) + LPV/RTV
Number analyzed (Participants) | 343 | 345
percentage of participants
  TLOVR | 62.6 | 61.1
  Obs | 84.3 | 86.8
  M/D=F | 64.3 | 62.3

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies/mL at Week 96
Description: A blood sample was drawn to determine the amount of HIV-1 RNA virus in copies/mL at Week 96. The percentage of participants with HIV-1 RNA <50 copies/mL at Week 96 were tabulated by treatment arm with stratification by baseline HIV-1 RNA levels (<100,000 copies/mL and >=100,000 copies/mL).
Time Frame: Week 96
Population: The Intent-To-Treat-Exposed (ITT-E) population. The secondary analysis methods were M=F, switch included, TLOVR, Observed, and M/D=F.
Measure: Number; unit: percentage of participants
Arm/Group | Abacavir/Lamivudine (ABC/3TC) + Lopinavir/Ritonavir (LPV/RTV) | Tenofovir/Emtricitabine (TDF/FTC) + LPV/RTV
Number analyzed (Participants) | 343 | 345
percentage of participants
  M=F, Switch Included | 59.9 | 58.0
  TLOVR | 52.1 | 51.0
  Obs | 86.9 | 91.3
  M/D=F | 56.4 | 54.5

4. Secondary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies/mL at Weeks 48 and 96 in Participants With Baseline HIV-1 RNA <100,000 Copies/mL
Description: A blood sample was drawn to determine the amount of HIV-1 RNA virus in copies/mL at Weeks 48 and 96. The percentage of participants with HIV-1 RNA <50 copies/mL at Weeks 48 and 96 were tabulated by treatment arm in participants with baseline HIV-1 RNA <100,000 copies/mL.
Time Frame: Weeks 48 and 96
Population: The Intent-To-Treat-Exposed (ITT-E) population. The secondary analysis methods were missing=failure (M=F), switch included, TLOVR, Observed, and M/D=F
Measure: Number; unit: percentage of participants
Arm/Group | Abacavir/Lamivudine (ABC/3TC) + Lopinavir/Ritonavir (LPV/RTV) | Tenofovir/Emtricitabine (TDF/FTC) + LPV/RTV
Number analyzed (Participants) | 188 | 205
percentage of participants
  M=F, Switch Included, Week 48 | 71 | 69
  TLOVR, Week 48 | 67 | 62
  Obs, Week 48 | 89 | 88
  MD=F, Week 48 | 68 | 62
  M=F, Switch Included, Week 96 | 63 | 58
  TLOVR, Week 96 | 57 | 52
  Obs, Week 96 | 89 | 94
  MD=F, Week 96 | 59 | 54

5. Secondary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies/mL at Weeks 48 and 96 in Participants With Baseline HIV-1 RNA >=100,000 Copies/mL
Description: A blood sample was drawn to determine the amount of HIV-1 RNA virus in copies/mL at Week 48 and 96. The percentage of participants with HIV-1 RNA <50 copies/mL at Weeks 48 and 96 were tabulated by treatment arm in participants with baseline HIV-1 RNA >=100,000 copies/mL.
Time Frame: Weeks 48 and 96
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Abacavir/Lamivudine (ABC/3TC) + Lopinavir/Ritonavir (LPV/RTV) | Tenofovir/Emtricitabine (TDF/FTC) + LPV/RTV
Number analyzed (Participants) | 155 | 140
percentage of participants
  M=F, Switch Included, Week 48 | 63 | 65
  TLOVR, Week 48 | 57 | 60
  Obs, Week 48 | 78 | 86
  M/D=F, Week 48 | 59 | 62
  M=F, Switch Included, Week 96 | 56 | 58
  TLOVR, Week 96 | 46 | 51
  Obs, Week 96 | 84 | 88
  M/D=F, Week 96 | 54 | 55

6. Secondary Outcome: Percentage of Participants With HIV-1 RNA <400 Copies/mL at Weeks 48 and 96
Description: A blood sample was drawn to determine the amount of HIV-1 RNA virus in copies/mL at Week 48 and 96. The percentage of participants with HIV-1 RNA <400 copies/mL at Weeks 48 and 96 were tabulated by treatment arm with stratification by baseline HIV-1 RNA levels (<100,000 copies/mL and >=100,000 copies/mL).
Time Frame: Weeks 48 and 96
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Abacavir/Lamivudine (ABC/3TC) + Lopinavir/Ritonavir (LPV/RTV) | Tenofovir/Emtricitabine (TDF/FTC) + LPV/RTV
Number analyzed (Participants) | 343 | 345
percentage of participants
  M=F, Switch Included, Week 48 | 75.2 | 71.3
  TLOVR, Week 48 | 70.9 | 66.4
  Obs, Week 48 | 93.8 | 92.2
  M/D=F, Week 48 | 71.4 | 66.2
  M=F, Switch Included, Week 96 | 63.9 | 61.2
  TLOVR, Week 96 | 58.4 | 56.3
  Obs, Week 96 | 92.8 | 96.3
  M/D=F, Week 96 | 60.1 | 56.9

7. Secondary Outcome: Percentage of Participants With HIV-1 RNA <400 Copies/mL at Weeks 48 and 96 in Participants With Baseline HIV-1 RNA <100,000 Copies/mL
Description: A blood sample was drawn to determine the amount of HIV-1 RNA virus in copies/mL at Weeks 48 and 96. The percentage of participants with HIV-1 RNA <400 copies/mL at Weeks 48 and 96 were tabulated by treatment arm in participants with baseline HIV-1 RNA <100,000 copies/mL.
Time Frame: Weeks 48 and 96
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Abacavir/Lamivudine (ABC/3TC) + Lopinavir/Ritonavir (LPV/RTV) | Tenofovir/Emtricitabine (TDF/FTC) + LPV/RTV
Number analyzed (Participants) | 188 | 205
percentage of participants
  M=F, Switch Included, Week 48 | 76 | 71
  TLOVR, Week 48 | 72 | 66
  Obs, Week 48 | 94 | 91
  M/D=F, Week 48 | 72 | 65
  M=F, Switch Included, Week 96 | 65 | 60
  TLOVR, Week 96 | 60 | 55
  Obs, Week 96 | 92 | 97
  M/D=F, Week 96 | 61 | 56

8. Secondary Outcome: Percentage of Participants With HIV-1 RNA <400 Copies/mL at Weeks 48 and 96 in Participants With Baseline HIV-1 RNA >=100,000 Copies/mL
Description: A blood sample was drawn to determine the amount of HIV-1 RNA virus in copies/mL at Weeks 48 and 96. The percentage of participants with HIV-1 RNA <400 copies/mL at Weeks 48 and 96 were tabulated by treatment arm in participants with baseline HIV-1 RNA >=100,000 copies/mL.
Time Frame: Weeks 48 and 96
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Abacavir/Lamivudine (ABC/3TC) + Lopinavir/Ritonavir (LPV/RTV) | Tenofovir/Emtricitabine (TDF/FTC) + LPV/RTV
Number analyzed (Participants) | 155 | 140
percentage of participants
  M=F, Switch Included, Week 48 | 75 | 71
  TLOVR, Week 48 | 70 | 67
  Obs, Week 48 | 94 | 94
  M/D=F, Week 48 | 71 | 68
  M=F, Switch Included, Week 96 | 63 | 63
  TLOVR, Week 96 | 56 | 58
  Obs, Week 96 | 93 | 96
  M/D=F, Week 96 | 59 | 58

9. Secondary Outcome: Median Change From Baseline in HIV-1 RNA at Week 48 and 96
Description: A blood sample was drawn to determine the amount of HIV-1 RNA virus in copies/mL at Weeks 48 and 96. Change from baseline was defined as HIV-1 RNA level at Weeks 48 and 96 minus HIV-1 RNA level at baseline.
Time Frame: Weeks 48 and 96
Population: The Intent-To-Treat-Exposed (ITT-E) population, observed analysis.
Measure: Median (Full Range); unit: log10 copies/mL
Arm/Group | Abacavir/Lamivudine (ABC/3TC) + Lopinavir/Ritonavir (LPV/RTV) | Tenofovir/Emtricitabine (TDF/FTC) + LPV/RTV
Number analyzed (Participants) | 236 | 219
log10 copies/mL
  Week 48 | -3.142 [-4.847 to 0.970] | -3.131 [-4.874 to 2.530]
  Week 96 | -3.114 [-5.304 to 0.819] | -3.165 [-4.874 to 0.139]

10. Secondary Outcome: Median Change From Baseline in CD4+ Cells at Weeks 48 and 96
Description: A blood sample was drawn to determine the CD4+ cell count at Weeks 48 and 96. Change from baseline was defined as CD4+ cell count at week 96 minus CD4+ cell count at baseline.
Time Frame: Weeks 48 and 96
Population: The Intent-To-Treat-Exposed (ITT-E) population, observed analysis.
Measure: Median (Full Range); unit: cells per cmm
Arm/Group | Abacavir/Lamivudine (ABC/3TC) + Lopinavir/Ritonavir (LPV/RTV) | Tenofovir/Emtricitabine (TDF/FTC) + LPV/RTV
Number analyzed (Participants) | 234 | 218
cells per cmm
  Week 48 | 201.0 [-170 to 903] | 173.0 [-190 to 921]
  Week 96 | 250.0 [-226 to 1033] | 246.5 [-116 to 793]

11. Secondary Outcome: Number of Participants Who Meet the Protocol-defined Virologic Failure (PDVF) Criteria at Week 96
Description: The number of participants that failed to respond to therapy based on the protocol definition of virologic failure (PDVF) was tabulated. PDVF was defined as either no confirmed HIV-1 RNA <200 copies/mL or HIV-1 RNA rebound >= 200 copies/mL on two consecutive occasions.
Time Frame: Baseline to Week 96
Population: The Intent-To-Treat-Exposed (ITT-E) population
Measure: Number; unit: participants
Arm/Group | Abacavir/Lamivudine (ABC/3TC) + Lopinavir/Ritonavir (LPV/RTV) | Tenofovir/Emtricitabine (TDF/FTC) + LPV/RTV
Number analyzed (Participants) | 343 | 345
participants
  Protocol-defined virologic failure | 49 | 48
  Fail to confirm HIV-1 RNA <200 copies/mL by wk 24 | 21 | 24
  Confirmed HIV-1 RNA rebound to >= 200 copies/mL | 28 | 24
  Suspected HIV-1 RNA rebound to >= 200 copies/mL | 12 | 11

12. Secondary Outcome: Number of Confirmed Virologic Failure Participants Who Had Treatment-emergent Genotypic Resistance Through 96 Weeks
Description: A blood sample was drawn for participants failing to respond to therapy and the mutations present in the virus were identified. For each participant, the mutations found at the time of failure were compared with any mutations found in the blood sample at baseline. New mutations that developed at the time of failure was tabulated by drug class. NRTI, nucleoside reverse transcriptase inhibitor; NNRTI, non-nucleoside reverse transcriptase inhibitor; PI, protease inhibitor.
Time Frame: Baseline and time of virologic failure (up to Week 96)
Population: Participants in the Intent-To-Treat-Exposed (ITT-E) population who met the confirmed virologic failure criteria with paired baseline and virologic failure genotypic evaluations
Measure: Number; unit: participants
Arm/Group | Abacavir/Lamivudine (ABC/3TC) + Lopinavir/Ritonavir (LPV/RTV) | Tenofovir/Emtricitabine (TDF/FTC) + LPV/RTV
Number analyzed (Participants) | 45 | 41
participants
  No. with paired genotypes at baseline and wk 96 | 45 | 41
  Participants with treatment-emergent mutations | 18 | 22
  NRTI-associated mutations | 11 | 17
  NNRTI-associated mutations | 4 | 3
  PI-associated mutations | 11 | 7

13. Secondary Outcome: Number of Confirmed Virologic Failure Participants at Week 96 With Genotypic Resistance to Lamivudine (3TC) and Emtricitabine (FTC) and Had Phenotypic Reduced Susceptibility
Description: A blood sample was drawn for participants failing to respond to therapy and the mutations present in the virus were identified. New mutations that developed to the NRTI class at the time of failure that no longer responded to lamivudine or emtricitabine were tabulated by drug class.
Time Frame: Baseline and time of virologic failure (up to Week 96)
Population: Participants in the Intent-To-Treat-Exposed (ITT-E) population who met the confirmed virologic failure criteria and had the M184 mutations.
Measure: Number; unit: participants
Arm/Group | Abacavir/Lamivudine (ABC/3TC) + Lopinavir/Ritonavir (LPV/RTV) | Tenofovir/Emtricitabine (TDF/FTC) + LPV/RTV
Number analyzed (Participants) | 11 | 17
participants
  Resistance NRTI class (M184V, M/V,M/I,A/V,I,M/I/V) | 11 | 17
  Reduced pheno susceptibility to lamivudine/M184V | 4 | 9
  Reduced phen susceptibility to lamivudine/M184M/V | 3 | 0
  Reduced pheno susceptibility to lamivudine/M184M/I | 0 | 1
  Reduced pheno susceptibility to lamivudine/M184A/V | 0 | 1
  Reduced pheno susceptibility to lamivudine/M184I | 0 | 1
  Reduced pheno suscept. to lamivudine/M184M/I/V | 0 | 1
  Reduced pheno suscept. to emtricitabine/M184V | 4 | 9
  Reduced pheno suscept. to emtricitabine/M184M/V | 3 | 0
  Reduced pheno suscept. to emtricitabine/M184M/I | 0 | 1
  Reduced pheno suscept. to emtricitabine/M184A/V | 0 | 1
  Reduced pheno suscept. to emtricitabine/M184I | 0 | 1
  Reduced pheno suscept. to emtricitabine/M184M/I/V | 0 | 1

14. Secondary Outcome: Number of Participants Who Reported a Suspected Abacavir Hypersensitivity Reaction (ABC HSR) Reaction or Proximal Renal Tubule Dysfunction
Description: The number of participants that experienced symptoms of a suspected abacavir hypersensitivity reaction was tabulated. The number of participants that developed laboratory signs of proximal renal tubule dysfunction was tabulated.
Time Frame: Baseline through 96 weeks
Population: The Safety population which included all randomized participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Abacavir/Lamivudine (ABC/3TC) + Lopinavir/Ritonavir (LPV/RTV) | Tenofovir/Emtricitabine (TDF/FTC) + LPV/RTV
Number analyzed (Participants) | 343 | 345
participants
  Participants (Par.) with suspected ABC HSR | 14 | 3
  Mild or Grade 1 | 1 | 0
  Moderate or Grade 2 | 8 | 2
  Severe or Grade 3 | 4 | 1
  Not Applicable | 1 | 0
  Par. with proximal renal tubule dysfunction | 0 | 5

ADVERSE EVENTS:
Arm/Group | Abacavir/Lamivudine (ABC/3TC) + Lopinavir/Ritonavir (LPV/RTV) | Tenofovir/Emtricitabine (TDF/FTC) + LPV/RTV
Serious Adverse Events (participants affected / at risk) | 42 | 45
Other Adverse Events (participants affected / at risk) | 182 | 182
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Abacavir/Lamivudine (ABC/3TC) + Lopinavir/Ritonavir (LPV/RTV) | Tenofovir/Emtricitabine (TDF/FTC) + LPV/RTV
Pneumonia (Infections and infestations) | 3/343 | 4/345
Gastroenteritis (Infections and infestations) | 1/343 | 1/345
Meningitis cryptococcal (Infections and infestations) | 1/343 | 1/345
Mycobacterium avium complex infection (Infections and infestations) | 0/343 | 2/345
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1/343 | 1/345
Staphylococcal infection (Infections and infestations) | 1/343 | 1/345
Abscess (Infections and infestations) | 0/343 | 1/345
Abscess limb (Infections and infestations) | 1/343 | 0/345
Bronchitis (Infections and infestations) | 0/343 | 1/345
Cellulitis (Infections and infestations) | 0/343 | 1/345
Cryptococcal fungaemia (Infections and infestations) | 1/343 | 0/345
Encephalitis viral (Infections and infestations) | 0/343 | 1/345
Gastroenteritis viral (Infections and infestations) | 1/343 | 0/345
Helicobacter infection (Infections and infestations) | 0/343 | 1/345
Kidney infection (Infections and infestations) | 1/343 | 0/345
Meningitis viral (Infections and infestations) | 1/343 | 0/345
Perianal abscess (Infections and infestations) | 1/343 | 0/345
Perirectal abscess (Infections and infestations) | 0/343 | 1/345
Pharyngitis streptococcal (Infections and infestations) | 1/343 | 0/345
Pneumonia bacterial (Infections and infestations) | 0/343 | 1/345
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0/343 | 1/345
Sepsis (Infections and infestations) | 0/343 | 1/345
Staphylococcal bacteraemia (Infections and infestations) | 0/343 | 1/345
Tonsilitis streptococcal (Infections and infestations) | 1/343 | 0/345
Tuberculosis (Infections and infestations) | 1/343 | 0/345
Upper respiratory tract infection (Infections and infestations) | 0/343 | 1/345
Drug hypersensitivity (Immune system disorders) | 12/343 | 3/345
Hypersensitivity (Immune system disorders) | 2/343 | 0/345
Immune reconstitution syndrome (Immune system disorders) | 2/343 | 0/345
Haematemesis (Gastrointestinal disorders) | 1/343 | 1/345
Nausea (Gastrointestinal disorders) | 0/343 | 2/345
Ascites (Gastrointestinal disorders) | 0/343 | 1/345
Diarrhoea (Gastrointestinal disorders) | 0/343 | 1/345
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0/343 | 1/345
Haemorrhoids (Gastrointestinal disorders) | 1/343 | 0/345
Proctitis (Gastrointestinal disorders) | 1/343 | 0/345
Vomiting (Gastrointestinal disorders) | 0/343 | 1/345
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/343 | 0/345
Carcinoid tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/343 | 1/345
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/343 | 1/345
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/343 | 0/345
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/343 | 1/345
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/343 | 0/345
Transient ischaemic attack (Nervous system disorders) | 1/343 | 1/345
Balance disorder (Nervous system disorders) | 0/343 | 1/345
Brain mass (Nervous system disorders) | 1/343 | 0/345
Brain stem infarction (Nervous system disorders) | 0/343 | 1/345
Cerebrovascular accident (Nervous system disorders) | 0/343 | 1/345
Migraine (Nervous system disorders) | 0/343 | 1/345
Syncope (Nervous system disorders) | 0/343 | 1/345
Chest pain (General disorders) | 2/343 | 0/345
Pyrexia (General disorders) | 1/343 | 1/345
Death (General disorders) | 0/343 | 1/345
Gait disturbance (General disorders) | 1/343 | 0/345
Non-cardiac chest pain (General disorders) | 0/343 | 1/345
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1/343 | 2/345
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1/343 | 0/345
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1/343 | 0/345
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0/343 | 1/345
Dependence (Psychiatric disorders) | 0/343 | 1/345
Depression (Psychiatric disorders) | 1/343 | 0/345
Major depression (Psychiatric disorders) | 0/343 | 1/345
Mental status changes (Psychiatric disorders) | 0/343 | 1/345
Suicide attempt (Psychiatric disorders) | 0/343 | 1/345
Anaemia (Blood and lymphatic system disorders) | 2/343 | 2/345
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1/343 | 1/345
Back pain (Musculoskeletal and connective tissue disorders) | 0/343 | 1/345
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0/343 | 1/345
Tendon pain (Musculoskeletal and connective tissue disorders) | 1/343 | 0/345
Cardiac arrest (Cardiac disorders) | 0/343 | 1/345
Cardiac failure congestive (Cardiac disorders) | 0/343 | 1/345
Cardiopulmonary failure (Cardiac disorders) | 0/343 | 1/345
Cholecystitis acute (Hepatobiliary disorders) | 1/343 | 0/345
Hepatitic cirrhosis (Hepatobiliary disorders) | 0/343 | 1/345
Hepatosplenomegaly (Hepatobiliary disorders) | 0/343 | 1/345
Hepatotoxicity (Hepatobiliary disorders) | 1/343 | 0/345
Haematuria (Renal and urinary disorders) | 0/343 | 1/345
Renal failure (Renal and urinary disorders) | 0/343 | 1/345
Renal failure acute (Renal and urinary disorders) | 0/343 | 1/345
Deep vein thrombosis (Vascular disorders) | 0/343 | 2/345
Hypertension (Vascular disorders) | 0/343 | 1/345
Concussion (Injury, poisoning and procedural complications) | 0/343 | 1/345
Fall (Injury, poisoning and procedural complications) | 1/343 | 0/345
Head injury (Injury, poisoning and procedural complications) | 1/343 | 0/345
Laceration (Injury, poisoning and procedural complications) | 0/343 | 1/345
Adrenal insufficiency (Endocrine disorders) | 1/343 | 0/345
Diabetic retinopathy (Eye disorders) | 0/343 | 1/345
Creatinine renal clearance decreased (Investigations) | 0/343 | 1/345
Dehydration (Metabolism and nutrition disorders) | 1/343 | 0/345
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/343 | 1/345
Ecchymosis (Skin and subcutaneous tissue disorders) | 0/343 | 1/345
Debridement (Surgical and medical procedures) | 1/343 | 0/345
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Abacavir/Lamivudine (ABC/3TC) + Lopinavir/Ritonavir (LPV/RTV) | Tenofovir/Emtricitabine (TDF/FTC) + LPV/RTV
Diarrhoea (Gastrointestinal disorders) | 85/343 | 80/345
Nausea (Gastrointestinal disorders) | 33/343 | 28/345
Blood triglycerides increased (Investigations) | 31/343 | 26/345
Upper respiratory tract infection (Infections and infestations) | 25/343 | 31/345
Glomerular filtration rate decreased (Investigations) | 21/343 | 28/345
Depression (Psychiatric disorders) | 25/343 | 23/345
Headache (Nervous system disorders) | 25/343 | 23/345
Blood cholesterol increased (Investigations) | 27/343 | 20/345
Sinusitis (Infections and infestations) | 19/343 | 24/345
Vomiting (Gastrointestinal disorders) | 21/343 | 15/345
Fatigue (General disorders) | 21/343 | 13/345

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.